CLINICAL TRIAL: NCT01925599
Title: Identification of Germline BAP1 Mutation In Subjects With Choroidal Nevi or Uveal Melanoma
Brief Title: BAP1 Testing in Instance Choroidal Nevi or Uveal Melanoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Amy C Schefler, MD (Other)
Responsible Party: Sponsor-Investigator, Amy C Schefler, MD, Director of Ophthalmic Oncology, Greater Houston Retina Research
Organization: Greater Houston Retina Research (Other)
Other Study IDs: BAP101
Record Dates: First submitted 2013-08-15; First posted 2013-08-20 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Choroidal Nevi, Uveal Melanoma
Keywords: Nevus; Choroidal Melanoma; BAP1 mutation
MeSH Terms: conditions — Uveal Melanoma; Nevus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The BAP1 trial will examine the blood of patients diagnosed with choroidal nevi or uveal melanoma for a germline BAP1 mutation and other genetic markers associated with developing malignancy as well as additional sequencing of the uveal melanoma genome.

DETAILED DESCRIPTION:
A germline BAP1 mutation predisposes a person to developing uveal melanoma and other cancers. If a mutation is discovered, it changes the potential approach to managing the nevus. In the presence of a known genomic change associated with aggressive disease, closer follow up and more aggressive treatment could preserve the patient's vision and prevent micrometastatic spread. This new screening technique will be able to extend the length and quality of life of patients with more frequent targeted cancer screens.

ELIGIBILITY:
Inclusion Criteria:

any person with choroidal nevi

* Willingness to provide signed informed consent
* Age > 18 years
* Diagnosis of choroidal nevi or uveal melanoma

Threre are no exclusionary criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age > 18 years, diagnosed with choroidal nevi or uveal melanoma
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2013-07; Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Examine the rate of germline BAP1 mutations in young patients, diagnosed with choroidal nevi | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Amy C. Schefler, MD, Principal Investigator — Retina Consultants Houston
Locations (3):
- United States (3):
  - Retina Consultants of Houston, Houston, Texas
  - Retina Consultants of Houston, Katy, Texas
  - Retina Consultants of Houston, The Woodlands, Texas

REFERENCES:
- [Background] Singh AD, Turell ME, Topham AK. Uveal melanoma: trends in incidence, treatment, and survival. Ophthalmology. 2011 Sep;118(9):1881-5. doi: 10.1016/j.ophtha.2011.01.040. Epub 2011 Jun 24. PMID 21704381
- [Background] Singh AD, Kalyani P, Topham A. Estimating the risk of malignant transformation of a choroidal nevus. Ophthalmology. 2005 Oct;112(10):1784-9. doi: 10.1016/j.ophtha.2005.06.011. PMID 16154197
- [Background] Jensen DE, Rauscher FJ 3rd. Defining biochemical functions for the BRCA1 tumor suppressor protein: analysis of the BRCA1 binding protein BAP1. Cancer Lett. 1999 Sep;143 Suppl 1:S13-7. doi: 10.1016/s0304-3835(99)90004-6. No abstract available. PMID 10546591
- [Background] Ventii KH, Devi NS, Friedrich KL, Chernova TA, Tighiouart M, Van Meir EG, Wilkinson KD. BRCA1-associated protein-1 is a tumor suppressor that requires deubiquitinating activity and nuclear localization. Cancer Res. 2008 Sep 1;68(17):6953-62. doi: 10.1158/0008-5472.CAN-08-0365. PMID 18757409
- [Background] Matatall KA, Agapova OA, Onken MD, Worley LA, Bowcock AM, Harbour JW. BAP1 deficiency causes loss of melanocytic cell identity in uveal melanoma. BMC Cancer. 2013 Aug 5;13:371. doi: 10.1186/1471-2407-13-371. PMID 23915344
- [Background] Abdel-Rahman MH, Pilarski R, Cebulla CM, Massengill JB, Christopher BN, Boru G, Hovland P, Davidorf FH. Germline BAP1 mutation predisposes to uveal melanoma, lung adenocarcinoma, meningioma, and other cancers. J Med Genet. 2011 Dec;48(12):856-9. doi: 10.1136/jmedgenet-2011-100156. Epub 2011 Sep 22. PMID 21941004